CLINICAL TRIAL: NCT07095062
Title: Structural-Functional Connectome and High Density Electroencephalogram: Pilot Study in Patients With Friedreich's Ataxia.
Brief Title: Electroencephalogram in Patients With Friedreich's Ataxia for the Study of the Structural and Functional Connectome.
Acronym: CONNETTOMA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Eugenio Medea (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 233-24; ANV 2025-28 (Registry Identifier: Comitato Etico Territoriale Area Nord Veneto)
Record Dates: First submitted 2025-07-02; First posted 2025-07-31 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Friedreich's Ataxia; Motor Disorders
Keywords: Functional Connectivity; HD-EEG; FRDA; Connectome; Cognitive Functioning; Neurodegenerative Disease; Cerebellar Disorders; Neurophysiological Biomarkers; Friedreich Ataxia
MeSH Terms: conditions — Friedreich Ataxia; Motor Disorders; Neurodegenerative Diseases; Cerebellar Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with Friedreich's ataxia undergoing HD-EEG and neurofunctional rehabilitation. (Experimental): This arm includes patients with a confirmed genetic diagnosis of Friedreich's Ataxia (FRDA), aged between 8 and 60 years, with SARA scale scores below 30. Participants undergo high-density electroencephalogram (HD-EEG) recording under resting conditions and during a motor task, as well as a comprehensive neuropsychological and emotional assessment. All follow an intensive rehabilitation program lasting 3-4 weeks. HD-EEG recordings are repeated after treatment and one year later to assess longitudinal changes in functional connectivity and identify potential biomarkers associated with clinical progression.
  Interventions: Device: HD-EEG recordings, combined with cognitive and motor assessment

INTERVENTIONS:
Device: HD-EEG recordings, combined with cognitive and motor assessment — Participants will undergo high-density EEG (HD-EEG) recordings under two conditions: at rest and while performing an upper limb motor task. The data obtained will be used to reconstruct source cortical activity and derive patterns of functional connectivity, using advanced neurophysiological analysis techniques, including the Avalanche Transition Matrix (ATM). In addition, patients will complete a neuropsychological assessment and participate in an intensive multidisciplinary rehabilitation program lasting 3 to 4 weeks, depending on age. The intervention aims to assess changes in the functional organization of the brain before and after treatment, as well as one year later, in order to explore potential biomarkers of disease progression.

SUMMARY:
Prospective, exploratory, multicenter pilot study investigating the structural and functional connectome in patients with Friedreich's Ataxia (FRDA) using high-density electroencephalogram (HD-EEG). The aim is to identify neurophysiological biomarkers and analyze the relationship between cortical connectivity, cognitive functioning, and clinical severity, particularly in response to rehabilitation treatment.

DETAILED DESCRIPTION:
Friedreich's Ataxia (FRDA) is a progressive neurodegenerative disease caused by mutations in the FXN gene, resulting in a reduction in the mitochondrial protein frataxin and a dysfunction in iron homeostasis. In addition to motor and sensory impairments, FRDA also results in cognitive and emotional deficits. Pathophysiologically, it is associated with cerebellar degeneration and alterations in cerebello-cortical networks.

The present study proposes a novel HD-EEG-based approach to analyze brain activity at resting-state and during the performance of a motor task (task-based) in subjects with FRDA. Thirty patients with confirmed genetic diagnosis, age between 8 and 60 years, and SARA score <30 will be recruited. EEG recordings will be performed in resting condition and during an upper limb motor task.

In addition to neurophysiological measures, each participant will undergo a comprehensive neuropsychological evaluation, including memory, attention, language, visuospatial skills, praxis, executive functions, emotional and personality aspects. Connectivity data will be correlated with cognitive profiles and scores on the SARA and mFARS clinical scales.

ELIGIBILITY:
Inclusion criteria:

* age between 8 and 60 years;
* genetic diagnosis of FRDA: presence of guanine-adenine trinucleotide (GAA) expansion in the two alleles of the fratassin gene, GAA1 and GAA2;
* score on the Scale for the Assessment and Rating of Ataxia (SARA) < 30;
* ability to take part in a neuropsychological assessment in Italian.

Exclusion criteria:

* age different from the range 8-60 years;
* diagnosis of acquired ataxia or other genetic ataxias;
* SARA scale score ≥ 30;
* inability to take part in an Italian-language neuropsychological assessment

Ages: 8 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-07-07 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Connectivity profile derived from HD-EEG in subjects with FRDA. | From enrollment to the end of treatment at 3 to 4 weeks and after 1 year of follow-up
  Characterization of alterations in the connectome derived from the HD-EEG of subjects with FRDA compared with matched controls;
Functional activity derived from HD-EEG in subjects with FRDA. | From enrollment to the end of treatment at 3 to 4 weeks and after 1 year of follow-up
  Evaluation of functional connectivity as a biomarker in the evolution of FRDA

SECONDARY OUTCOMES:
Correlation between functional connectivity/activity and quantitative parameters derived from neuropsychological scales. Correlation between functional connectivity/activity and quantitative parameters derived from motor scales (SARA and mFARS). | From enrollment to the end of treatment at 3 to 4 weeks and after 1 year of follow-up
  1. acquisition of new knowledge about the neuronal basis of impaired neurocognitive functioning in FRDA;
  2. evaluation of possible correlations with disease severity scales pre- and post-rehabilitation treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Gabriella Paparella, Medical Doctor, Principal Investigator — IRCCS E. Medea / Associazione la Nostra Famiglia
Locations (1):
- IRCCS Eugenio Medea / Associazione la Nostra Famiglia, Conegliano, Treviso, Italy

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual participant data will be shared with other researchers upon reasonable request
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Start date: January 2028 End date: January 2038
Access Criteria: Any researchers accredited by non-profit clinical and research center